CLINICAL TRIAL: NCT06457295
Title: Impact of Diabetes Mellitus on Retinal Microvasculature in Patients Without Clinical Retinopathy Using Optical Coherence Tomography Angiography
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdou Saeed, principal investigator, Sohag University
Other Study IDs: Soh-Med-24-05-16MS
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Retinopathy, DR
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- non-diabetic: patients who are above 40 years old and don't have diabetes
  Interventions: Diagnostic Test: optical coherence tomography angiography
- diabetic (0-5y): patients who are above 40 years old and have diabetes for less than 5 years
  Interventions: Diagnostic Test: optical coherence tomography angiography
- diabetics (5-10y): patients who are above 40 years old and have diabetes for 5-10 years
  Interventions: Diagnostic Test: optical coherence tomography angiography
- diabetics (10y < ): patients who are above 40 years old and have diabetes for more than 10 years
  Interventions: Diagnostic Test: optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: optical coherence tomography angiography — A non-invasive eye imaging technique that creates high-resolution, 3D maps of blood flow in the retina and choroid by comparing sequential OCT scans to detect the motion of red blood cells to provide a visual contrast to the static tissue that allows the visualization the retinal microvasculature without needing an injectable dye, unlike traditional angiography.

SUMMARY:
the aim of this study is to assess the impact of duration of DM on OCTA parameters in diabetic patients without clinical Diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Type of DM: Type 2.
2. Fundus examination: no macular edema or other signs of clinical retinopathy

Exclusion Criteria:

1. Ocular history : any history of significant ocular injury or disease that could affect the retinal microvasculature such as retinal vascular occlusion, glaucoma, or vitreo-macular disease, as such conditions have also been noted to show sub-clinical OCTA changes [13, 14].
2. Fundus examination: macular edema or any other signs of clinical retinopathy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients will be recruited from diabetics who will present for retinopathy screening examination at outpatient clinic of Sohag University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
FAZ metrics | baseline
  FAZ area, FAZ perimeter & FAZ flow density
Superficial Vessel Density | baseline
  foveal, average parafoveal & average perifoveal
Deep Vessel Density | baseline
  foveal, average parafoveal, average perifoveal
SCP thickness | baseline
  foveal, average parafoveal & average perifoveal
DCP thickness | baseline
  foveal, average parafoveal & average perifoveal
Sectoral superficial vessel density | baseline
  superior parafoveal, inferior parafoveal, nasal parafoveal, temporal parafoveal, superior perifoveal, inferior perifoveal, nasal perifoveal & temporal perifoveal
Sectoral deep vessel density | baseline
  superior parafoveal, inferior parafoveal, nasal parafoveal, temporal parafoveal, superior perifoveal, inferior perifoveal, nasal perifoveal & temporal perifoveal

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rao HL, Pradhan ZS, Suh MH, Moghimi S, Mansouri K, Weinreb RN. Optical Coherence Tomography Angiography in Glaucoma. J Glaucoma. 2020 Apr;29(4):312-321. doi: 10.1097/IJG.0000000000001463. PMID 32053551

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT06457295/Prot_SAP_000.pdf